CLINICAL TRIAL: NCT00529399
Title: Effects of Recombinant Human Glutamic Acid Decarboxylase (rhGAD65) Formulated in Alum (GAD-alum) on the Progression of Type 1 Diabetes in New Onset Subjects
Brief Title: Effects of Recombinant Human Glutamic Acid Decarboxylase on the Progression of Type 1 Diabetes in New Onset Subjects
Acronym: TN08
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Center for Research Resources (NCRR) (NIH); American Diabetes Association (Other); Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TN08 GAD65; U01DK061055 (NIH); UC4DK097835 (NIH)
Record Dates: First submitted 2007-09-12; First posted 2007-09-14 (Estimated); Results first posted 2016-12-07 (Estimated); Last update posted 2020-05-07 (Actual); Status verified 2020-04

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: immune tolerance; immunotherapy; antigen-specific tolerance; vaccine induced tolerance; Beta-cell function; T-cells; DPT-1; treatment of type 1 diabetes; new onset type 1 diabetes; juvenile diabetes; T1D; diabetes mellitus; Type 1 diabetes TrialNet; TrialNet
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — Aluminum Hydroxide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 1 (Experimental): 3 injections of GAD-Alum vaccine
  Interventions: Drug: GAD-Alum
- 2 (Experimental): 2 injections of GAD-Alum vaccine and one injection with Aluminum hydroxide alone
  Interventions: Drug: GAD-Alum and Aluminum hydroxide
- 3 (Placebo Comparator): 3 injections of Aluminum hydroxide alone
  Interventions: Drug: Aluminum hydroxide

INTERVENTIONS:
Drug: GAD-Alum — Participants will receive 3 injections of 20 micrograms GAD-Alum subcutaneously. The first two injections are given 4 weeks apart and the second and third are given 8 weeks apart.
  Other Names: Diamyd
  Arms: 1
Drug: GAD-Alum and Aluminum hydroxide — Participants will receive 3 injections subcutaneously. The first two will contain 20 micrograms GAD-Alum vaccine and are given 4 weeks apart. The third injection will be Aluminum hydroxide alone and will be given 8 weeks after the second injection.
  Other Names: Diamyd
  Arms: 2
Drug: Aluminum hydroxide — Participants will receive 3 injections of Aluminum hydroxide alone, subcutaneously. The first two injections are given 4 weeks apart and the second and third are given 8 weeks apart.
  Other Names: Alhydrogel
  Arms: 3

SUMMARY:
The purpose of this study is to determine whether treatment with multiple injections of GAD-Alum will preserve the body's own (endogenous) insulin production in patients who have been recently diagnosed with type 1 diabetes mellitus (T1DM).

DETAILED DESCRIPTION:
Type 1 diabetes (T1D) is an autoimmune disease. This means that the immune system (the part of the body which helps fight infections) mistakenly attacks and destroys the cells that produce insulin (islet cells found in the pancreas called islet cells). As these cells are destroyed, the body's ability to produce insulin decreases. Glutamic acid decarboxylase (GAD) is one of the major autoantigens (a protein that the immune system is reacting to) involved in the autoimmune process underlying T1DM.

GAD-Alum is Recombinant human (rhGAD65) and is used as an antigen-specific immune modulator. Previous studies have shown that it may slow or prevent autoimmune destruction of pancreatic islet cells by introducing "immune tolerance". By administering excess autoantigen, the body may stop its attack on its own cells that produce insulin. If the immune system's attack can be halted in a patient with recent onset T1DM, than residual insulin secretion may be maintained. This may be beneficial in decreasing acute and long-term diabetic complications as well as improving glucose control.

ELIGIBILITY:
Inclusion Criteria:

* Age 3 to 45 years - Insulin dependent type 1-diabetes mellitus diagnosed within the previous 3 months
* Stimulated C-peptide levels greater than or equal to 0.2 pmol/ml measured during a mixed meal tolerance test (MMTT) conducted 3 weeks from diagnosis of diabetes
* Presence of GAD65 antibodies
* At least one month from last immunization
* Willing to comply with intensive diabetes management
* If participant is a woman with reproductive potential, she must be willing to avoid pregnancy and have a negative pregnancy test
* Willing to forgo routine clinical immunizations during the first 100 days after initial study drug administration

Exclusion Criteria:

* Immunodeficiency or clinically significant chronic lymphopenia
* Active infection
* Positive PPD test result
* Pregnant or lactating or anticipating becoming pregnant for 24 months following first injection
* Ongoing use of medications known to influence glucose tolerance
* Require use of systemic immunosuppressant(s)
* Serologic evidence of current or past HIV, Hep B, or Hep C infection
* History of malignancies
* Ongoing use of non-insulin pharmaceuticals to affect glycemic control
* Participation in another clinical trial with a new chemical entity within the past 3 months
* Complicating medical issues or abnormal clinical laboratory results that interfere with study conduct or cause increased risk including neurological, or clinically significant blood count abnormalities (such as lymphopenia, leukopenia, or thrombocytopenia)
* History of epilepsy, head trauma or cerebrovascular accident or clinical
* History of alcohol or drug abuse

Ages: 3 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 145 (Actual)
Dates: Start 2009-02; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diane Wherrett, M.D., Principal Investigator — University of Toronto, Hospital for Sick Children; Jay Skyler, M.D., Study Chair — University of Miami
Locations (15):
- United States (14):
  - Childrens Hospital of Los Angeles, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of California-San Francisco, San Francisco, California
  - Barbara Davis Center for Childhood Diabetes/University of Colorado Health Sciences Center, Aurora, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - University of Miami/ Miller School of Medicine, Miami, Florida
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Joslin Diabetes Center, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Columbia University, New York, New York
  - Childrens Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas/Southwestern Medical School, Dallas, Texas
  - Benaroya Research Institute, Seattle, Washington
- Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data are available at the NIDDK Central Repository: https://repository.niddk.nih.gov/studies/tn08-gad-new-onset/?query=tn08
URL: https://repository.niddk.nih.gov/studies/tn08-gad-new-onset/?query=tn08

REFERENCES:
- [Background] Atkinson MA, Eisenbarth GS. Type 1 diabetes: new perspectives on disease pathogenesis and treatment. Lancet. 2001 Jul 21;358(9277):221-9. doi: 10.1016/S0140-6736(01)05415-0. PMID 11476858
- [Background] Pleau JM, Fernandez-Saravia F, Esling A, Homo-Delarche F, Dardenne M. Prevention of autoimmune diabetes in nonobese diabetic female mice by treatment with recombinant glutamic acid decarboxylase (GAD 65). Clin Immunol Immunopathol. 1995 Jul;76(1 Pt 1):90-5. doi: 10.1006/clin.1995.1092. PMID 7606872
- [Background] Tian J, Clare-Salzler M, Herschenfeld A, Middleton B, Newman D, Mueller R, Arita S, Evans C, Atkinson MA, Mullen Y, Sarvetnick N, Tobin AJ, Lehmann PV, Kaufman DL. Modulating autoimmune responses to GAD inhibits disease progression and prolongs islet graft survival in diabetes-prone mice. Nat Med. 1996 Dec;2(12):1348-53. doi: 10.1038/nm1296-1348. PMID 8946834
- [Background] Tisch R, Liblau RS, Yang XD, Liblau P, McDevitt HO. Induction of GAD65-specific regulatory T-cells inhibits ongoing autoimmune diabetes in nonobese diabetic mice. Diabetes. 1998 Jun;47(6):894-9. doi: 10.2337/diabetes.47.6.894. PMID 9604865
- [Background] Tisch R, Wang B, Weaver DJ, Liu B, Bui T, Arthos J, Serreze DV. Antigen-specific mediated suppression of beta cell autoimmunity by plasmid DNA vaccination. J Immunol. 2001 Feb 1;166(3):2122-32. doi: 10.4049/jimmunol.166.3.2122. PMID 11160264
- [Background] Jun HS, Chung YH, Han J, Kim A, Yoo SS, Sherwin RS, Yoon JW. Prevention of autoimmune diabetes by immunogene therapy using recombinant vaccinia virus expressing glutamic acid decarboxylase. Diabetologia. 2002 May;45(5):668-76. doi: 10.1007/s00125-002-0806-9. Epub 2002 Apr 4. PMID 12107747
- [Result] Wherrett DK, Bundy B, Becker DJ, DiMeglio LA, Gitelman SE, Goland R, Gottlieb PA, Greenbaum CJ, Herold KC, Marks JB, Monzavi R, Moran A, Orban T, Palmer JP, Raskin P, Rodriguez H, Schatz D, Wilson DM, Krischer JP, Skyler JS; Type 1 Diabetes TrialNet GAD Study Group. Antigen-based therapy with glutamic acid decarboxylase (GAD) vaccine in patients with recent-onset type 1 diabetes: a randomised double-blind trial. Lancet. 2011 Jul 23;378(9788):319-27. doi: 10.1016/S0140-6736(11)60895-7. Epub 2011 Jun 27. PMID 21714999
- See also: Related Info — http://www.diabetestrialnet.org/
- See also: Related Info — http://www.jdrf.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The original recruitment goal was to enroll 126 subjects. However, additional eligible subjects were identified during the screening process and 145 subjects were enrolled in the study.
Groups:
- GAD-alum: 3 injections of Glutamic Acid Decarboxylase (GAD)-Alum vaccine
  GAD-Alum: Participants will receive 3 injections of 20 micrograms GAD-Alum subcutaneously. The first two injections are given 4 weeks apart and the second and third are given 8 weeks apart.
- GAD-alum Plus Alum: 2 injections of GAD-Alum vaccine and one injection with Aluminum hydroxide alone
  GAD-Alum: Participants will receive 3 injections subcutaneously. The first two will contain 20 micrograms GAD-Alum vaccine and are given 4 weeks apart. The third injection will be Aluminum hydroxide alone and will be given 8 weeks after the second injection.
- Alum Alone: 3 injections of Aluminum hydroxide alone
  Aluminum hydroxide: Participants will receive 3 injections of Aluminum hydroxide alone, subcutaneously. The first two injections are given 4 weeks apart and the second and third are given 8 weeks apart.
Period: Overall Study
Arm/Group | GAD-alum | GAD-alum Plus Alum | Alum Alone
Started | 48 | 49 | 48
Completed | 46 | 48 | 46
Not Completed | 2 | 1 | 2
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Non-compliant | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- GAD-alum: 3 injections of GAD-Alum vaccine
  GAD-Alum: Participants will receive 3 injections of 20 micrograms GAD-Alum subcutaneously. The first two injections are given 4 weeks apart and the second and third are given 8 weeks apart.
- Total: Total of all reporting groups
Arm/Group | GAD-alum | GAD-alum Plus Alum | Alum Alone | Total
Number analyzed (Participants) | 48 | 49 | 48 | 145
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.8 (10.3) | 14.8 (8.7) | 16.6 (9.2) | 16.4 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 31 | 19 | 64
  Male | 34 | 18 | 29 | 81

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome is the Area Under the Stimulated C-peptide Curve (AUC) at the One Year Visit
Description: The primary outcome is the area under the stimulated C-peptide curve (AUC) based on data collected at time 0 to 2 hours of a 4-hour mixed meal glucose tolerance test (MMTT) conducted at the primary endpoint visit. The timed measurements are done at: 0, 15, 30 60, 90, and 120 minutes.
Time Frame: Based on mixed meal tolerance test (MMTT) conducted at the one year visit
Measure: Geometric Mean (95% Confidence Interval); unit: nmol/L
Arm/Group | GAD-alum | GAD-alum Plus Alum | Alum Alone
Number analyzed (Participants) | 46 | 48 | 46
nmol/L | 0.448 [0.361 to 0.540] | 0.350 [0.267 to 0.438] | 0.418 [0.333 to 0.508]
Statistical Analysis 1: Comparison: GAD-alum vs Alum Alone; The calculation for the concentration of c-peptide is a weighted average of the 6 timed measurements of c-peptide in nano-moles/Liter. We try to distinguish this calculation from the AUC by referring to it as the "AUC mean" and may be expressed algebraically as the AUC/(120 min.); thus, the units are the same as the y-axis; Test type: Superiority or Other; p = 0.98, ANCOVA
Statistical Analysis 2: Comparison: GAD-alum Plus Alum vs Alum Alone; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.51, ANCOVA

ADVERSE EVENTS:
Arm/Group | GAD-alum | GAD-alum Plus Alum | Alum Alone
Serious Adverse Events (participants affected / at risk) | 5/48 | 3/49 | 5/48
Other Adverse Events (participants affected / at risk) | 20/48 | 25/49 | 24/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GAD-alum (N=48) | GAD-alum Plus Alum (N=49) | Alum Alone (N=48)
Cardiac ischemia/infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Endocrine - Other (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Infection - Other (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Lymphatics - Other (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Neurology - Other (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Personality/behavioral (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Intra-operative Injury - Other (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GAD-alum (N=48) | GAD-alum Plus Alum (N=49) | Alum Alone (N=48)
Auditory/Ear- Other (Ear and labyrinth disorders) | 0 (0) | 3 (3) | 0 (0)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0)
Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 4 (8) | 7 (13) | 0 (0)
Endocrine - Other (Endocrine disorders) | 0 (0) | 3 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (3)
Infection - Other (Infections and infestations) | 10 (14) | 10 (13) | 10 (16)
Sinus Infection with unknown ANC (Infections and infestations) | 3 (4) | 0 (0) | 0 (0)
Musculoskeletal/Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (6) | 10 (10)
Pain- Abdomen NOS (General disorders) | 0 (0) | 3 (3) | 0 (0)
Pain - Other (General disorders) | 0 (0) | 0 (0) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (9) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No